CLINICAL TRIAL: NCT03576196
Title: Preoperative Pain Neuroscience Education Combined With Therapeutic Exercise Post-surgery in Patients With Carpal Tunnel Syndrome. A Double-blind Randomized Controlled Trial
Brief Title: Preoperative Pain Neuroscience Education in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clínico La Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNC-001
Record Dates: First submitted 2018-05-14; First posted 2018-07-03 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: physical therapy; Pain; disability; kinesiophobia.
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (Experimental): Single session of pain neuroscience education a week prior to surgery, of an individual character, lasting approximately 30 minutes, performed by a physiotherapist trained. The main contents addressed in the educational session were: neurophysiological aspects of pain, biopsychosocial aspects of pain, concept of peripheral and central sensitization, using audio-visual support, examples and metaphors for a better understanding by the patient, as reported in previous studies.
  This treatment was combined with a hand therapy session seven days after the surgery, verbal and written instruction was given to the patients to perform exercises at home of active sliding of the digital flexor tendon, active opposition of the thumb and active range of flexion and extension of the wrist.
  Interventions: Other: Preoperative Pain Neuroscience Education
- Usual Care (Other): Patients in the control group received "usual care", which consists of an educational session prior to surgery, based on medical, anatomical and pathological aspects of the syndrome.
  This treatment was combined with a hand therapy session seven days after the surgery, verbal and written instruction was given to the patients to perform exercises at home of active sliding of the digital flexor tendon, active opposition of the thumb and active range of flexion and extension of the wrist.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Preoperative Pain Neuroscience Education — Single session of pain neuroscience education a week prior to surgery, of an individual character, lasting approximately 30 minutes, performed by a physiotherapist trained. The main contents addressed in the educational session were: neurophysiological aspects of pain, biopsychosocial aspects of pain, concept of peripheral and central sensitization, using audio-visual support, examples and metaphors for a better understanding by the patient, as reported in previous studies.
  This treatment was combined with a hand therapy session seven days after the surgery, verbal and written instruction was given to the patients to perform exercises at home of active sliding of the digital flexor tendon, active opposition of the thumb and active range of flexion and extension of the wrist.
  Other Names: Experimental
  Arms: Pain Neuroscience Education
Other: Usual Care — This treatment was combined with a hand therapy session seven days after the surgery, verbal and written instruction was given to the patients to perform exercises at home of active sliding of the digital flexor tendon, active opposition of the thumb and active range of flexion and extension of the wrist.
  Other Names: Control
  Arms: Usual Care

SUMMARY:
Study Design: A double-blind randomized controlled study.

Background: Patients operated on for carpal tunnel release surgery may persist with pain after surgery, which could be modulated by psychosocial factors such as depression, catastrophic thinking and kinesiophobia.

Objectives: To evaluate the efficacy of a preoperative session in pain neuroscience education combined with postoperative therapeutic exercise in the perception of pain, functionality and psychosocial variables in patients following carpal tunnel release.

Methods: Thirty participants were randomly assigned to the pain neuroscience education group combined with postoperative therapeutic exercise (n = 15) or to the control group with preoperative usual care combined with postoperative therapeutic exercise (n = 15). Evaluations included the Visual Analogue Scale (VAS), Disability of Arm, Shoulder, and Hand Questionnaire (QuickDASH), pain Catastrophizing Scale (PCS), Tampa scale of kinesiophobia (TSK-11) and Hospital Anxiety and Depression Scale (HADS) . A basal, fourth and twelfth week measurement was made.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Medical diagnosis of Carpal Tunnel Syndrome waiting for surgery
* Agree to participate in the study.

Exclusion Criteria:

* Inability to understand instructions,
* Illiteracy,
* Previous participation in educational programs regarding pain,
* Pathology of uncontrolled mental health,
* Cognitive problems,
* Previous surgeries in the operated extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Change of Disability in upper-limb | Change from Baseline Disability at fourth and twelfth week
  The Perception of patients of their disability in upper-limb evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH) Spanish version Outcome Measure is a 30-item scored 1-5. The assigned values for all completed responses are simply summed and averaged. Scoring: The assigned values for all completed responses are simply summed and averaged and higher values represent a worse Disability in upper-limb.

SECONDARY OUTCOMES:
Change of Pain Interference: Kinesiophobia | Change from Baseline Kinesiophobia at fourth and twelfth week
  Kinesiophobia will be evaluated by Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
Change of Emotional status: Hospital Anxiety and Depression Scale (HAD). | Change from Baseline emotional status at fourth and twelfth week
  Patient's emotional state will be evaluated by Hospital Anxiety and Depression Scale (HAD), which assess the level of anxiety and depression. Subscales and score range are Anxiety (0-21) and Depression (0-21). Scoring: items of each subscale are summed, indicating: 0-7 normality, 8-10 probably case, 11-21 anxiety or depression clinical case. Higher values represent a worse outcome.
Change of Pain evaluation: | Change from Baseline Pain at fourth and twelfth week
  Pain will be measured by the Visual Analog Scale for pain (VAS) from 0 to 10, where higher values represent a worse outcome (0 is no pain and 10 the maximum pain experienced).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico La Florida, Santiago, RM, Chile